CLINICAL TRIAL: NCT06181747
Title: Research on the Development of Attention and Its Relationship With Emotions in Children and Adolescents
Brief Title: Development of Attention and Its Relationship With Emotions in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Psychology, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2KM011639-K12023000015
Record Dates: First submitted 2023-12-01; First posted 2023-12-26 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD group (Experimental): Participants are required to engage in game training at home for 5 days per week, with each session lasting 20-25 minutes. The game is equipped with anti-addiction measures, limiting the maximum daily game time to 30 minutes. Participants will adjust their game training based on their own abilities, and as the training progresses, the game will adaptively adjust the difficulty level and change levels accordingly.
  Interventions: Device: a serious mobile device-based game prototype (Save the Muse Home)
- healthy control group (Experimental): Participants are required to engage in game training at home for 5 days per week, with each session lasting 20-25 minutes. The game is equipped with anti-addiction measures, limiting the maximum daily game time to 30 minutes. Participants will adjust their game training based on their own abilities, and as the training progresses, the game will adaptively adjust the difficulty level and change levels accordingly.
  Interventions: Device: a serious mobile device-based game prototype (Save the Muse Home)

INTERVENTIONS:
Device: a serious mobile device-based game prototype (Save the Muse Home) — The cognitive impairment corresponding to the symptoms, which we are interested in, focuses on executive inhibition, motor inhibition, sustained attention, selective attention, working memory, and planning ability. The training content will be presented in different scenarios as effective training components. The story line of the warrior breakthrough runs through the whole game, each level is adapted according to the functional damage areas of different patients, and each level involves reward and punishment mechanisms to keep the interest of the players, the difficulty gradient of each level is kept moderate, and the game includes design elements such as space, time, object attributes, actions, rules, skills, and probabilities, etc., which ultimately completes Save the Muse Home, a serious game for the treatment of ADHD.

SUMMARY:
Our aim was to describe the development and usability of a mobile device-based game therapy software for ADHD.

DETAILED DESCRIPTION:
A total of 51 ADHD children and 52 healthy children were included in the study. At baseline, subjects underwent tests such as ADHD symptom-related scale assessments, computer-assisted information processing tests, and physiological-psychological tests, after which participants completed a 4-week game intervention training at home. After complete completion of the intervention, subjects repeated all tests from the baseline period and answered treatment satisfaction questions.

ELIGIBILITY:
Inclusion Criteria:

* ADHD-a. Age between 6-12 years, any gender.
* ADHD-b. Outpatient patients diagnosed with ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
* ADHD-c. Patients and/or their guardians willing to participate in the study and provide informed consent. Participants aged 8 and above should also sign a child's informed consent form.
* HC. The control group of healthy participants are recruited from a secondary school in Nanjing, matching the age and gender of the ADHD group.

Exclusion Criteria:

* a. Neurodevelopmental disorders such as cerebral palsy, epilepsy, adrenoleukodystrophy, and other similar conditions.
* b. Severe mental disorders including tic disorders, autism spectrum disorders, intellectual disability, schizophrenia, bipolar disorder, depressive disorders, specific learning disorders, and other significant psychiatric conditions.
* c. Individuals exhibiting ADHD-like symptoms due to hearing impairments.
* d. Requirement of any central nervous system medication (including both traditional and Western medicine as well as dietary supplements) such as antipsychotics or antidepressants at any stage of the study.
* e. Patients who have received systematic treatment with two different categories of ADHD medications without improvement.
* f. Individuals with color blindness or any other condition that would prevent proper use of the software.
* g. History of or current gaming addiction.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Continuous Performance Test, CPT | baseline and post (an average of 30days after baseline)
  CPT software is one of the commonly used tools for examining attention and is a computer-assisted information processing test with objective results, independent of supervisors, and is the most widely used experimental paradigm in current research. The CPT paradigm adopted in this study is the presence of a white boxed area on a black background on the calculator screen, with white squares randomly appearing above or below the white boxed area, requiring the target stimulus to be a right mouse button press when the square appears below it.

SECONDARY OUTCOMES:
Swanson Nolan, and Pelham-IV rating scales, SNAP-IV | baseline and post (an average of 30days after baseline)
  The SNAP-IV rating scales (Swanson Nolan, and Pelham-IV rating scales, SNAP-IV) is a revised version of the Swanson, Nolan Pelham (SNAP) (Swanson, et al., 1983), which was developed based on the description of ADHD symptoms in the Diagnostic and Statistical Manual of Mental Disorders (DSM). It consists of three subscales: attention deficit, hyperactivity-impulsivity, and oppositional defiance, and is mainly used for screening, diagnostic support, and assessment of treatment efficacy and symptom improvement in children and adolescents between the ages of 6 and 18 years. Although SNAP-IV consists of 3 subscales, it is one scale, just like SDQ and BRIEF mentioned later.
Strengths and Difficulties Questionnaire, SDQ | baseline and post (an average of 30days after baseline)
  The SDQ is a brief behavioral screening questionnaire designed and developed by American psychologist Goodman R in 1997 based on the Diagnostic and Statistical Manual of Mental Disorders-IV and the Diagnostic Criteria for the Classification of Mental and Behavioral Disorders, 10th Edition (ICD-10). It is used to assess behavioral and emotional problems in children and adolescents and has good reliability and validity.
Behavior Rating Inventory of Executive Function, BRIEF | baseline and post (an average of 30days after baseline)
  The scale consists of 86 entries in two major areas: the Behavior Management Index (BMI), which includes the three subscales of Inhibition, Conversion, and Affect, and Control, Conversion and Affect, and Control subscales; and the Metacognitive Functioning Index: five subscales including Task Initiation, Working Memory, Planning, Organization, and Monitoring. It has good reliability and validity.
Anti-saccade task | baseline and post (an average of 30days after baseline)
  First, present the central gaze point cross for 2s, the central cross disappeared while the target appeared as a green dot, randomly present four positions at 3°, 6° left and right sides horizontally, presentation time 1000ms, each angle randomly appeared 5 times for a total of 20 times, when the response is over a 300ms feedback point will appear in the correct position.
Delay-saccade task | baseline and post (an average of 30days after baseline)
  Presentation of the central gaze point cross for 2 s, the target stimulus appeared (the cross continued to exist) for the green origin randomly presented at four positions 3°, 6° left and right sides horizontally, presentation time 100 ms. Subsequently, the gaze point was presented only at the center of the screen for 1, 3, and 5 s, staring at the cross intently, and then the screen appeared to go blank for 1.4 s, the subject recalled looking at the beginning of the target, and the latter a 200-ms feedback point appeared at the correct location.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengkui Liu, Ph.D., Principal Investigator — Institute of Psychology, Chinese Academy of Sciences
Locations (2):
- China (2):
  - Nanjing Normal University, Nanjing, Jiangsu
  - Institute of Psychology, Chinese Academy of Sciences, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo J, Li F, Wu Y, Liu X, Zheng Q, Qi Y, Huang H, Xu G, Liu Z, He F, Zheng Y. A mobile device-based game prototype for ADHD: development and preliminary feasibility testing. Transl Psychiatry. 2024 Jun 10;14(1):251. doi: 10.1038/s41398-024-02964-2. PMID 38858375